CLINICAL TRIAL: NCT01909778
Title: An Open Label Single Dose Phase I Trial of 120 mg and 240 mg BI 201335 Soft Gel Capsules to Study Pharmacokinetic Properties and Safety in Patients With Compensated Liver Cirrhosis in Historical Comparison With 1220.2
Brief Title: Open Label Single Dose Phase I Trial of BI 201335 to Study Pharmacokinetics and Safety in Patients With Compensated Liver Cirrhosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1220.15; 2007-007776-42 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-07-25; First posted 2013-07-29 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Hepatitis C; Liver Cirrhosis
MeSH Terms: conditions — Hepatitis C; Liver Cirrhosis | interventions — faldaprevir

ARMS (1):
- BI 201335 (Experimental): BI 201335 two single oral doses, separated by 14 days washout period
  Interventions: Drug: BI 201335

INTERVENTIONS:
Drug: BI 201335 — single oral doses

SUMMARY:
This trial was intended to investigate the pharmacokinetics, safety and tolerability of BI 201335 NA soft-gel capsules in patients with compensated liver cirrhosis, i.e. grade A according to Child-Pugh classification (< 7 points).

ELIGIBILITY:
Inclusion criteria:

1. Patients with liver cirrhosis, that is histologically proven in a previous liver biopsy; possible aetiologies are: cured HCV infection, former alcohol abuse, genetic haemochromatosis, non-alcoholic steatohepatitis or others.
2. Compensated liver disease, as indicated by Prothrombin time or INR prolonged to <1.7 x ULN, serum bilirubin < 2 mg/dl, albumin > 3.5 g/dl, no ascites or encephalopathy (Child-Pugh grade A, score < 7)
3. Age 18 years or older
4. Male patients, or female with documented hysterectomy, ovariectomy or tubal ligation OR menopausal female with last menstrual period at least 12 months prior to screening OR female of childbearing potential with a negative serum pregnancy test at screening and day 1 and willing to ensure consistent and correct contraception
5. Written informed consent prior to study enrolment which must be consistent with international conference on harmonisation ¿ good clinical practice (ICH-GCP) and local legislation.

Exclusion criteria:

1. Serological evidence of active HBV, HCV or HIV infection (i.e. seropositivity for HBs antigen, anti-HIV-1 or -2 antibodies; if anti-HCV antibody positive, patients must have documented negative HCV RNA for at least 12 months)
2. Usage of any drug within 7 days or 5 halftimes, whichever is longer, prior to treatment; or the planned usage of a drug during the course of the current study
3. Usage of any investigational drug within 30 days prior to treatment; or the planned usage of an investigational drug during the course of the current study
4. Decompensated liver disease within past 12 months, as indicated by variceal bleeding, ascites, encephalopathy, Prothrombin time or INR prolonged to > 1,7 x ULN, serum bilirubin > 2 mg/dl or albumin < 3,5 g/dl (i.e. Child-Pugh grade B)
5. ALT or AST levels > 5xULN, Alkaline Phosphatase > 2xULN
6. Liver cirrhosis due to primary or secondary biliary cirrhosis, sclerosing cholangitis, vanishing bile duct disease
7. History of alcohol abuse within the past 3 months
8. Known hypersensitivity to any content of the study drug
9. Pregnant or breast feeding females
10. Females of childbearing potential who are not willing to ensure consistent and correct use of condoms and at least one additional medically accepted method of contraception (diaphragm with spermicidal substance, cervical caps) or who are unwilling to comply to complete abstinence, from the date of screening until 6 months after the last dose of study drug
11. AFP value > 100 ng/ml; if AFP is > 20 and <= 100 ng/ml, patients can be included if liver cancer is excluded by two congruent imaging studies (i.e. ultrasound plus CT scan or MRI)
12. Evidence of chronic kidney failure (i.e. serum creatinine > ULN)
13. Haemoglobinopathy (e.g., thalassaemia major or sickle cell anaemia)
14. Concomitant intercurrent illnesses including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness or social situation that would limit compliance with trial requirement or which are considered relevant for the evaluation of the pharmacokinetic parameters or safety of the trial drug.
15. Active or suspected malignancy or history of malignancy within the last 2 years (with the exception of appropriately treated basal cell carcinoma or in situ carcinoma of the uterine cervix)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1220.15.49006 Boehringer Ingelheim Investigational Site, Mainz, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects: The trial was a nonrandomised, open-label, 2-period fixed-sequence trial to evaluate two single oral doses of Faldaprevir, separated by 14 days washout period. The dose levels were 120 mg first, 240 mg second.
  A number of 12 entered patients with compensated liver cirrhosis was planned.
Period: Overall Study
Arm/Group | All Subjects
Started | 2
Completed | 1
Not Completed | 1
Not completed — failed screening | 1

BASELINE CHARACTERISTICS:
Population: While a number of 12 entered patients with non-HCV liver cirrhosis was planned, only a total of 2 patients were enrolled in 1 centre in Germany.
Groups:
- All Subjects: The trial was a nonrandomised, open-label, 2-period fixed-sequence trial to evaluate two single oral doses of Faldaprevir, separated by 14 days washout period. The dose levels were 120 mg and 240 mg.
  A number of 12 entered patients with compensated liver cirrhosis was planned.
Arm/Group | All Subjects
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: AUC 0-∞
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC 0-∞).
Time Frame: -0:15, 1:00, 2:00, 3:00, 4:00, 5:00, 6:00, 8:00, 12:00, 16:00, 20:00, 24:00, 48:00, 72:00, 96:00, 120:00 h (hours) after drug administration on day 1 and day 15
Population: Only one patient was treated and completed this study; he was the only patient analysed.
Measure: Number; unit: h*ng/mL
Groups:
- Low Dose of Faldaprevir (Period 1): single dose of 120 mg Faldaprevir soft gel capsule.
- High Dose of Faldaprevir (Period 2): single dose of 240 mg Faldaprevir soft gel capsule after a wash-out period of at least 14 days.
Arm/Group | Low Dose of Faldaprevir (Period 1) | High Dose of Faldaprevir (Period 2)
Number analyzed (Participants) | 1 | 1
h*ng/mL | 7240 | 24700

2. Primary Outcome: Cmax
Description: Maximum plasma concentration (Cmax). Individual Cmax values will be directly determined from the plasma concentration time profiles.
Time Frame: -0:15, 1:00, 2:00, 3:00, 4:00, 5:00, 6:00, 8:00, 12:00, 16:00, 20:00, 24:00, 48:00, 72:00, 96:00, 120:00 h after drug administration on day 1 and day 15
Population: Only one patient was treated and completed this study; he was the only patient analysed.
Measure: Number; unit: ng/mL
Arm/Group | Low Dose of Faldaprevir (Period 1) | High Dose of Faldaprevir (Period 2)
Number analyzed (Participants) | 1 | 1
ng/mL | 308 | 999

3. Secondary Outcome: Tmax
Description: Time at which the maximum plasma concentration occurs (tmax). Individual tmax values will be directly determined from the plasma concentration time profiles.
Time Frame: as for outcome 2
Population: Only one patient was treated and completed this study; he was the only patient analysed.
Measure: Number; unit: hours
Arm/Group | Low Dose of Faldaprevir (Period 1) | High Dose of Faldaprevir (Period 2)
Number analyzed (Participants) | 1 | 1
hours | 8.00 | 8.00

4. Secondary Outcome: AUC0-tz
Description: Area under the concentration-time curve over the time interval from 0 to the last quantifiable plasma concentration (AUC0-tz).
Time Frame: as for outcome 2
Population: Only one patient was treated and completed this study; he was the only patient analysed.
Measure: Number; unit: h*ng/mL
Arm/Group | Low Dose of Faldaprevir (Period 1) | High Dose of Faldaprevir (Period 2)
Number analyzed (Participants) | 1 | 1
h*ng/mL | 6770 | 23900

5. Secondary Outcome: t1/2
Description: Elimination half-life (t1/2). The terminal half-life will be calculated from the terminal rate constant.
Time Frame: as for outcome 2
Population: Only one patient was treated and completed this study; he was the only patient analysed.
Measure: Number; unit: hours
Arm/Group | Low Dose of Faldaprevir (Period 1) | High Dose of Faldaprevir (Period 2)
Number analyzed (Participants) | 1 | 1
hours | 33.8 | 26.8

6. Secondary Outcome: CL/F
Description: Apparent clearance of the analyte in plasma following extravascular administration (CL/F).
  The apparent clearance after oral administration will be determined according to the following equation: CL or CL/F=dose/AUC0-∞. (F=absolute bioavailability factor)
Time Frame: as for outcome 2
Population: Only one patient was treated and completed this study; he was the only patient analysed.
Measure: Number; unit: mL/min
Arm/Group | Low Dose of Faldaprevir (Period 1) | High Dose of Faldaprevir (Period 2)
Number analyzed (Participants) | 1 | 1
mL/min | 276 | 162

7. Secondary Outcome: Vz/F
Description: Apparent volume of distribution during the terminal phase (Vz/F) following an extravascular dose (at steady state).
Time Frame: as for outcome 2
Population: Only one patient was treated and completed this study; he was the only patient analysed.
Measure: Number; unit: Liter
Arm/Group | Low Dose of Faldaprevir (Period 1) | High Dose of Faldaprevir (Period 2)
Number analyzed (Participants) | 1 | 1
Liter | 809 | 376

8. Secondary Outcome: MRTpo
Description: Mean residence time of the analyte in the body after oral administration (MRTpo).
Time Frame: as for outcome 2
Population: Only one patient was treated and completed this study; he was the only patient analysed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Low Dose of Faldaprevir (Period 1) | High Dose of Faldaprevir (Period 2)
Number analyzed (Participants) | 1 | 1
hours | 39.3 (NA) — Not calculable as only one participant analysed. | 31.6 (NA) — Not calculable as only one participant analysed.

9. Secondary Outcome: Assessment of Tolerability by Investigator
Description: The investigator has assessed tolerability based on adverse events and the laboratory evaluation. Tolerability was assessed by the investigator according to the categories 1="good", 2="satisfactory", 3="not satisfactory", and 4="bad".
Time Frame: Day 6 of period 1 and 2
Population: Only one patient was treated and completed this study; he was the only patient analysed.
Measure: Number; unit: units on a scale
Arm/Group | Low Dose of Faldaprevir (Period 1) | High Dose of Faldaprevir (Period 2)
Number analyzed (Participants) | 1 | 1
units on a scale | 1 | 1

10. Secondary Outcome: Clinical Relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinanalysis and ECG
Description: Clinical Relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinanalysis and ECG. New abnormal findings or worsening of baseline conditions were reported as Adverse Events.
Time Frame: from intake of the second dose Faldaprevir up to 9 days
Population: Only one patient was treated and completed this study; he was the only patient analyzed.
Measure: Number; unit: participants
Arm/Group | Low Dose of Faldaprevir (Period 1) | High Dose of Faldaprevir (Period 2)
Number analyzed (Participants) | 1 | 1
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From intake of the second dose Faldaprevir up to 9 days. Patients were required to report spontaneously any adverse events (AEs) as well as the time of onset, duration and intensity of these events.
Description: In addition, each patient was assessed by an investigator at any measurement time point as well as at the end of observation and whenever necessary as deemed by the investigator. Assessment was made using non-specific questions such as "How do you feel?". Specific questions were asked wherever required or useful to more precisely describe an AE.
Arm/Group | Low Dose of Faldaprevir (Period 1) | High Dose of Faldaprevir (Period 2)
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose of Faldaprevir (Period 1) (N=1) | High Dose of Faldaprevir (Period 2) (N=1)
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1
Sweating (Skin and subcutaneous tissue disorders) | 0 | 1
Soft stools (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.